CLINICAL TRIAL: NCT06629506
Title: Prospective Evaluation of MicroMatrix® Flex in Wounds Complicated by Tunneling and Undermining
Brief Title: MicroMatrix® Flex in Tunneling Wounds
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-MMFLEX-001
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pressure Injury; Venous Ulcer; Necrotizing Soft Tissue Infection; Diabetic Ulcers; Draining Wound
MeSH Terms: conditions — Pressure Ulcer; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects with tunneling and/or undermining wounds (Experimental): MicroMatrix Flex, MicroMatrix UBM Particulate, and Cytal Wound Matrix 2-Layer will be used to treat the wound.
  Interventions: Device: MicroMatrix® Flex; Device: MicroMatrix® UBM Particulate; Device: Cytal® Wound Matrix 2-Layer

INTERVENTIONS:
Device: MicroMatrix® Flex — MicroMatrix® Flex is intended for the management of wounds including: partial and full-thickness wounds, pressure ulcers, venous ulcers, diabetic ulcers, chronic vascular ulcers, tunneled/undermined wounds, surgical wounds (donor sites/grafts, post-Mohs surgery, post-laser surgery, podiatric, wound dehiscence), trauma wounds (abrasions, lacerations, partial thickness burns, skin tears), draining wounds. The device is intended for one-time use.
Device: MicroMatrix® UBM Particulate — MicroMatrix® UBM Particulate is intended for the management of wounds including: partial and full-thickness wounds, pressure ulcers, venous ulcers, diabetic ulcers, chronic vascular ulcers, tunneled/undermined wounds, surgical wounds (donor sites/grafts, post-Moh's surgery, post-laser surgery, podiatric, wound dehiscence), trauma wounds (abrasions, lacerations, second-degree burns, skin tears), and draining wounds. The device is intended for one-time use.
Device: Cytal® Wound Matrix 2-Layer — Cytal® Wound Matrix is intended for the management of wounds including: partial and full-thickness wounds, pressure ulcers, venous ulcers, diabetic ulcers, chronic vascular ulcers, tunneled/undermined wounds, surgical wounds (donor sites/grafts, post-Moh's surgery, post-laser surgery, podiatric, wound dehiscence), trauma wounds (abrasions, lacerations, second-degree burns, skin tears), and draining wounds. The device is intended for one-time use.

SUMMARY:
To evaluate the safety and performance of MicroMatrix® Flex in subjects with wounds complicated by tunneling and/or undermining features.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and performance of MicroMatrix® Flex in subjects with wounds complicated by tunneling and/or undermining features. Prospective data will be collected to assess the rate of wound area/volume reduction (progression toward closure) and post-operative complications at 12 weeks, and rate of skin graft take, when applicable, up to 16 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 22 years at the time of consent
2. Patient with a diagnosis of pressure injury, venous ulcer, diabetic ulcer, necrotizing soft tissue infection associated wound, dehiscing and/or draining wounds associated with open abdominal procedures, or any indication per the Instructions For Use
3. Patient is willing and able to adhere to protocol requirements and comply with the study follow-up regimen
4. Patient has reviewed the IRB/IEC-approved consent form, has been properly consented per the protocol and has documented their consent to participate in the study by signing the IRB/IEC-approved consent form

Exclusion Criteria:

1. Burn as etiology of wound
2. Unmanaged infection and/or osteomyelitis as determined pre-operatively
3. Known allergy, hypersensitivity, or objection to porcine materials, due to religion, culture, or other
4. Patient report of concurrent participation in another clinical trial that would interfere with this study
5. Any condition, concomitant medication, or concomitant treatment that, in the opinion of the investigator, would preclude the use of the study device or preclude the patient from completing the follow-up requirements

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Relative rate of closure of a tunneling or undermining feature | At 12 weeks or skin graft visit
  Relative rate of closure of a tunneling or undermining feature as determined manually, through measurement of opening size and depth of managed wound at 12 weeks or skin graft visit, relative to first visit/application post debridement

SECONDARY OUTCOMES:
Relative rate of closure of a tunneling or undermining feature | First device application through to 12 weeks
  Relative rate of closure of a tunneling or undermining feature as determined manually, through measurement of opening size and depth of managed wound at each visit, relative to first visit/application post debridement
Relative rate of overall wound closure | First device application through to 12 weeks
  Relative rate of overall wound closure as determined manually, through measurement of volume, using the Kundin method, of managed wound at each visit, relative to first visit/application post debridement
Relative rate of overall wound closure | First device application through to 12 weeks
  Relative rate of overall wound closure per number of treatments received
Number of wound infections, seromas, and hematomas | First device application through to 12 weeks
  Number of wound infections, seromas, and hematomas requiring re-intervention (including incision and drainage)
Number of managed wounds which require removal of devices | First device application through to 12 weeks
  Number of managed wounds which require removal of devices due to complications, allergic reactions, or intolerance of devices
Length of stay in-patient | First device application through to 12 weeks
  Length of stay in-patient, if applicable

OTHER OUTCOMES:
Area of skin graft | At skin graft visit, a maximum of 14 weeks from first device application
  Area of skin graft utilized relative to the original wound size
Skin graft take | At skin graft visit + (4 weeks ± 7 days)
  Skin graft take percentage at skin graft follow-up
Time to graft | First device application through to skin graft visit
  Time to skin graft

CONTACTS AND LOCATIONS:
Overall Officials: Claire Witherel, Ph.D., Study Director — Integra LifeSciences Corporation
Locations (3):
- United States (3):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - MedStar Health Research Institute Inc., Washington D.C., District of Columbia
  - Northwell Comprehensive Wound Healing Center, Lake Success, New York

IPD SHARING:
Plan to Share IPD: No